CLINICAL TRIAL: NCT00171743
Title: Switch From Tacrolimus to Cyclosporine Microemulsion: Immunosuppressive Agents and Diabetes Management in Liver Transplant Recipients in Maintenance (DIALIVER)
Brief Title: Efficacy and Safety of Cyclosporine Microemulsion in Diabetic Adult Stable Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceticals
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: COLO400AIT03
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Liver Transplant
Keywords: Adults; Post transplant diabetes

INTERVENTIONS:
Drug: Cyclosporine microemulsion

SUMMARY:
The purpose of this study is to determine whether the switch from tacrolimus to cyclosporine microemulsion benefits post-transplant diabetes management (in terms of glycogenic control and insulin dosage) in stable liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 months post-transplant
* Patients in treatment with tacrolimus
* Post-transplant diabetes treated with insulin for at least one month

Exclusion Criteria

* Known hypersensitivity to cyclosporine microemulsion
* Investigational drug within 60 days before baseline or during the study
* Patients who cannot comply with the study requirements

Other protocol-defined exclusion criteria applied

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-04; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Rathi M, Rajkumar V, Rao N, Sharma A, Kumar S, Ramachandran R, Kumar V, Kohli HS, Gupta KL, Sakhuja V. Conversion from tacrolimus to cyclosporine in patients with new-onset diabetes after renal transplant: an open-label randomized prospective pilot study. Transplant Proc. 2015 May;47(4):1158-61. doi: 10.1016/j.transproceed.2014.12.050. PMID 26036543